CLINICAL TRIAL: NCT03598647
Title: Affective Responses to Physical Activity: A Novel Intervention Target for Increasing Physical Activity
Brief Title: Feelings About Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1179772
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2019-11

CONDITIONS: Physical Activity; Obesity
Keywords: exercise; physical activity; obesity; weight loss
MeSH Terms: conditions — Motor Activity; Obesity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical activity information - for non-exercisers only (Active Comparator): Non-exercisers randomized to this condition will receive basic information about physical activity. This includes the national physical activity guidelines,clarification of 'moderate-intensity', exercise safety, and the progression of physical activity within the weight loss program.
  Interventions: Behavioral: Physical activity information
- Affect and physical activity - for non-exercisers only (Experimental): Non-exercisers randomized to this condition will receive the same basic information about physical activity as described above, but they will also receive a brief intervention focused on affective responses to exercise.
  Interventions: Behavioral: Affect and physical activity
- Exercisers (No Intervention): Engaging in >=150 min/week of moderate-intensity exercise over the past 6 months and a most recent typical week
- Non-exercisers (No Intervention): Engaging in <30 min/week of moderate-intensity exercise over the past 6 months and a most recent typical week

INTERVENTIONS:
Behavioral: Affect and physical activity — The focus of this intervention is to help the participant to become more aware of their positive feelings and experiences related to exercise. They will learn about typical affective responses to exercise, view their own affective responses to exercise, and they will be taught cognitive strategies for altering affective responses to exercise. Participants will also receive general information about exercise safety, physical activity guidelines, and exercise intensity.
  Arms: Affect and physical activity - for non-exercisers only
Behavioral: Physical activity information — Participants will receive general information about exercise safety, physical activity guidelines, and exercise intensity.
  Arms: Physical activity information - for non-exercisers only

SUMMARY:
This study seeks to investigate why some individuals exercise more than others by focusing on feelings related to exercise. This two part study first examines whether regular exercisers (n=30) and non-exercisers (n=30) differ in how a 30-minute moderate-intensity exercise bout makes them feel. All participants will walk on a treadmill for 30 minutes on two separate occasions and will be asked to report on how they feel before, during, and after exercise, how they anticipate that exercise will make them feel, and how they remembered feeling during exercise. In addition, after exercise session #2, non-exercisers will be randomized to: 1) a brief intervention focused on providing general information about the physical activity guidelines, or 2) a brief intervention which provides general information about physical activity guidelines, but also focuses on affective responses to physical activity. Non-exercisers will complete an identical, third exercise session approximately 1-week following this intervention. Further, all participants will receive a 12-week, Internet-delivered weight loss program following all exercise visits and physical activity will be assessed before and after the weight loss program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* BMI between 25.0 and <40.0 kg/m2
* Either a 'Non-exerciser', defined as reporting exercising at a moderate-intensity for <30 min/week over the past 6 months and a most recent typical week or an 'exerciser', defined as exercising for ≥150 min/week over the past 6 months and a most recent typical week.

Exclusion Criteria:

* Presence of any condition that would limit one's ability to exercise (e.g., orthopedic limitations)
* History of coronary artery disease (i.e., myocardial infarction or symptoms of angina), stroke, diabetes, or pulmonary disease (e.g., COPD or emphysema).
* Currently taking any medication that would alter heart rate (e.g., beta blocker)
* Women who are pregnant or nursing
* Uncontrolled hypertension (resting blood pressure ≥140/90 mmHg)
* Exercising >30 min/week but <150 min/week (i.e., neither 'non-exerciser' nor 'exerciser')
* Use of medications for weight loss, or current participation in another weight loss program
* Bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Unick, PhD, Principal Investigator — The Miriam Hospital; Kathryn Demos, PhD, Principal Investigator — The Miriam Hospital; David Williams, PhD, Principal Investigator — Brown University
Locations (1):
- Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity Information: After the completion of exercise sessions 1 and 2 (which were necessary for the aims comparing exercisers vs. non-exercisers), non-exercisers randomized to this condition received basic information about physical activity, including the national physical activity guidelines, clarification of 'moderate-intensity', exercise safety, and the progression of physical activity within the weight loss program.
- Affect and Physical Activity: After the completion of exercise sessions 1 and 2 (which were necessary for the aims comparing exercisers vs. non-exercisers), non-exercisers randomized to this condition received the same basic information about physical activity as the 'physical activity information' group but they also received a brief intervention focused on affective responses to exercise. The focus of this intervention was to help the participant to become more aware of their positive feelings and experiences related to exercise. They learned about typical affective responses to exercise, viewed their own affective responses to exercise, and were taught cognitive strategies for altering affective responses to exercise.
Period: Exercisers vs. Non-exercisers
Arm/Group | Exercisers | Non-exercisers | Physical Activity Information | Affect and Physical Activity
Started | 30 | 30 | 0 | 0
Completed | 29 | 30 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Period: Interventions for Non-exercisers
Arm/Group | Exercisers | Non-exercisers | Physical Activity Information | Affect and Physical Activity
Started | 0 | 0 | 14 | 16
Completed | 0 | 0 | 14 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercisers | Non-exercisers | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (8.9) | 45.0 (11.3) | 47.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 30 | 59
Self-reported exercise minutes (min/week) over past 6 months [Mean (Standard Deviation); unit: min/week] | 285.9 (148.8) | 14.0 (15.2) | 147.6 (172.0)

OUTCOME MEASURES:

1. Primary Outcome: Pre-exercise Affect (Session 1)
Description: Measured using Feeling Scale (FS) prior to exercise bout. Scores range from -5 to +5 with higher values indicating more positive affect
Time Frame: Prior to exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercisers | Non-exercisers
Number analyzed (Participants) | 29 | 30
units on a scale | 3.97 (1.40) | 2.70 (2.15)

2. Primary Outcome: Mean During Exercise Affect (Session 1)
Description: Average during exercise Feeling Scale (FS) score which was assessed every 5 minutes during exercise. Feeling Scale scores range from -5 to +5 with higher values indicating more positive affect.
Time Frame: average score assessed every 5 minutes during exercise, up to 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercisers | Non-exercisers
Number analyzed (Participants) | 29 | 30
units on a scale | 3.53 (1.64) | 2.71 (1.54)

3. Primary Outcome: Post-exercise Affect (Session 1)
Description: Feeling Scale (FS) score 15 minutes post-exercise. Feeling Scale scores range from -5 to +5 with higher values indicating more positive affect.
Time Frame: 15 minutes post-exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercisers | Non-exercisers
Number analyzed (Participants) | 29 | 30
units on a scale | 4.03 (1.32) | 3.80 (1.27)

4. Primary Outcome: Memory of During Exercise Affect (Session 1) - Calculated as the Difference Between Recalled During Exercise Affect and Actual During Exercise Affect
Description: Calculated as follows: recalled during exercise affect (assessed 7 days post-exercise) minus actual during exercise affect (average of Feeling Scale scores every 5 minutes during exercise). Possible scores for both recalled affect and actual affect range from -5 to +5, where higher numbers indicate more positive affect. A negative change value indicates that participants remembered feeling less positive during exercise than they actually felt.
Time Frame: average score assessed every 5 minutes during exercise, up to 30 minutes, and 7 days post-exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercisers | Non-exercisers
Number analyzed (Participants) | 29 | 30
units on a scale | -.77 (1.22) | -.80 (1.23)

5. Primary Outcome: Memory of Post-exercise Affect (Session 1) - Calculated as the Difference Between Recalled Post-exercise Affect and Actual Post-exercise Affect
Description: Calculated as follows: recalled post-exercise affect (assessed 7 days following exercise session) minus actual post-exercise affect (Feeling Scale score assessed 15 minutes post-exercise). Possible scores for both recalled affect and actual affect range from -5 to +5, where higher numbers indicate more positive affect. A negative change value indicates that participants remembered feeling less positive post-exercise than they actually felt.
Time Frame: 15 minutes and 7 days post-exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercisers | Non-exercisers
Number analyzed (Participants) | 29 | 30
units on a scale | -1.07 (1.21) | -0.76 (1.81)

6. Primary Outcome: Anticipated During Exercise Affect (Session 2)
Description: How one anticipates that they will feel during exercise session 2 (an exercise session that is identical to exercise session 1).This was assessed prior to exercise session 2 via a 100 mm visual analogue scale (range 1-100) where a higher number indicates more positive affect.
Time Frame: prior to exercise session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercisers | Non-exercisers
Number analyzed (Participants) | 29 | 30
units on a scale | 71.3 (18.7) | 54.1 (21.3)

7. Secondary Outcome: Pre-exercise Affect (Session 3)
Description: as for outcome 1
Time Frame: Prior to exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Physical Activity Information: Non-exercisers randomized to this condition will receive basic information about physical activity. This includes the national physical activity guidelines,clarification of 'moderate-intensity', exercise safety, and the progression of physical activity within the weight loss program.
  Physical activity information: Participants will receive general information about exercise safety, physical activity guidelines, and exercise intensity.
- Affect and Physical Activity: Non-exercisers randomized to this condition will receive the same basic information about physical activity as described above, but they will also receive a brief intervention focused on affective responses to exercise.
  Affect and physical activity: The focus of this intervention is to help the participant to become more aware of their positive feelings and experiences related to exercise. They will learn about typical affective responses to exercise, view their own affective responses to exercise, and they will be taught cognitive strategies for altering affective responses to exercise. Participants will also receive general information about exercise safety, physical activity guidelines, and exercise intensity.
Arm/Group | Physical Activity Information | Affect and Physical Activity
Number analyzed (Participants) | 14 | 16
units on a scale | 2.11 (1.70) | 2.94 (1.53)

8. Secondary Outcome: Mean During Exercise Affect (Session 3)
Description: as for outcome 2
Time Frame: average score assessed every 5 minutes during exercise, up to 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity Information | Affect and Physical Activity
Number analyzed (Participants) | 14 | 16
units on a scale | 3.14 (1.69) | 3.14 (1.24)

9. Secondary Outcome: Post-exercise Affect (Session 3)
Description: as for outcome 3
Time Frame: 15 minutes post-exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity Information | Affect and Physical Activity
Number analyzed (Participants) | 14 | 16
units on a scale | 3.71 (1.27) | 3.94 (0.85)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Physical Activity Information: Non-exercisers randomized to this condition will receive basic information about physical activity. This includes the national physical activity guidelines, clarification of 'moderate-intensity', exercise safety, and the progression of physical activity within the weight loss program.
  Physical activity information: Participants will receive general information about exercise safety, physical activity guidelines, and exercise intensity.
Arm/Group | Exercisers | Non-exercisers | Physical Activity Information | Affect and Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03598647/Prot_001.pdf
  • Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT03598647/SAP_002.pdf
  • Informed Consent Form (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03598647/ICF_000.pdf